CLINICAL TRIAL: NCT02176707
Title: Modelling of Quality Life, Clinical and Physiological Measures in Idiopathic Pulmonary Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of East Anglia (Other)
Collaborators: InterMune (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014RESP03L; 14/SW/0047 (Other Grant/Funding Number: InterMune)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Idiopathic Pulmonary Fibrosis; Dyspnoea; Anxiety; Depression
Keywords: Lung Function; Exercise Capacity
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Dyspnea; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Idiopathic pulmonary fibrosis sufferers

SUMMARY:
As there are no validated tools for assessing patient reported outcomes or health related quality of life in idiopathic pulmonary fibrosis (IPF), different studies have utilised different methods. This means that comparison of the outcomes of studies is difficult or inaccurate. By collecting different quality of life tools and patient reported outcome at the same time, it will be possible to map or model the results of one tool or groups of tools onto another. 250 patients with IPF will be asked to complete the EuroQoL 5D, Kings Brief Interstitial Lung Disease questionnaire, St George's Respiratory Questionnaire, MRC dyspnoea scale, University of California, San Diego shortness of breath questionnaire and the Hospital Anxiety and Depression Scale, along with spirometry every 3 months, and undergo a 6 minute walk test every 6 months, over a 12 month period. Prognostic models will be constructed from all the clinical (questionnaire and function) measures a linear regression model.

DETAILED DESCRIPTION:
There are no validated or accepted tools for assessing health related quality of life (HRQOL) or dyspnoea in patients with idiopathic pulmonary fibrosis (IPF) and there are no accepted or recommended tools for assessing patient reported outcomes in clinical trials of patients with IPF. Assessment of these outcomes is important to patients and may be considered the most crucial outcome measures of an intervention in IPF. With this in mind, the majority of the recently reported randomised clinical studies in IPF have evaluated HRQOL and dyspnoea, most commonly as secondary outcomes, but this has been achieved by different tools. For example the Capacity studies(1) utilised the St George's Respiratory Questionnaire whereas the ASCEND (Efficacy and Safety of Pirfenidone in Patients With Idiopathic Pulmonary Fibrosis) (http://clinicaltrial.gov/ct2/show/NCT01366209) study is currently assessing dyspnoea using the University of California, San Diego shortness of breath questionnaire. As there is no method of directly comparing HRQOL between different clinical evaluations in IPF, there is a desperate need to produce algorithms for relating the different outcome measures in IPF.

The St George's Respiratory Questionnaire(2) is the most commonly utilised tool in trials of IPF(3-5). Although it relates to physiological impairment in IPF(6), it was developed in patients with Chronic Obstructive Pulmonary Disease (COPD) and therefore lacks content validity. An abbreviated version (SGRQ-I) containing the questions most relevant to IPF has therefore been developed and validated(7). The Kings Brief Interstitial Lung disease (K-BILD) questionnaire is a recently validated tool for patients with interstitial lung disease not specifically idiopathic pulmonary fibrosis(8) but has not been utilised in multicentre studies to measure treatment interventions in IPF. The EuroQol 5D (EQ5D) is a well-validated global health status instrument designed for use in clinical and health-economic trials(9). This has been validated in chronic respiratory disease and has been used in several studies(4, 5, 10). In terms of assessing dyspnoea, studies have utilised the University of California, San Diego (UCSD) shortness of breath questionnaire (SOBQ)(4, 11), the medicine research council (MRC) dyspnoea score(5), and the transition dyspnoea index(12).

The investigators have conducted a brief mapping exercise based on the data from patients randomised to the placebo arm of the Treating idiopathic pulmonary fibrosis with the addition of co-trimoxazole (TIPAC) study(5). The SGRQ data were mapped onto the EQ5D data using pairs of data from individuals at the same time point with the addition demographic and lung function data(unpublished). This mapping exercise produced an equation with greater predictive strength than using data from COPD patients showing that modelling algorithms are disease specific information cannot be shared between different respiratory conditions. The investigators now wish to undertake a larger study to generate more accurate models to approximate the EQ5D and also to explore the relationship between other patient reported outcome measures. It is only by undertaking this work, that the results of individual studies can be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 40 years.
* IPF based on multi-disciplinary following review of clinical history, thoracic high resolution computed tomography (HRCT) and/or usual interstitial pneumonia (UIP) histology confirmed by surgical lung biopsy consensus according to international guidelines.
* Patients may receive oral prednisolone up to a dose of 10 mg per day, anti-oxidant therapy or pirfenidone at study entry.

Exclusion Criteria:

* A recognised significant co-existing respiratory disease, defined as a respiratory condition that exhibits a clinically relevant effect on respiratory symptoms and disease progression as determined by the principal investigator following multi-disciplinary discussion. For example, patients with bronchiectasis will only be included if the bronchiectasis is deemed to be traction bronchiectasis as a result of idiopathic pulmonary fibrosis.
* Airflow obstruction defined as a FEV1/FVC<60% predicted or a residual volume greater than 120% predicted.
* Significant medical, surgical or psychiatric disease that in the opinion of the patient's attending physician would exhibit a clinically relevant effect on the patient's health related quality of life.
* Unable to provide written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by hospital databases, patient registries and clinical notes and approached by the patients' attending physician or clinical team.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
St George's Respiratory Questionnaire (SGRQ) | 12 month period
  St George's Respiratory Questionnaire (SGRQ) is a tool for assessing quality of life that has previously been validated for the use with patients with interstitial lung disease. It is a responsive tool that has three domains: symptoms, activity and impact (on daily life)
Kings Brief Interstitial Lung Disease questionnaire (K-BILD) | 12 month period
  Kings Brief Interstitial Lung Disease questionnaire (K-BILD) Recently developed, this is a disease specific questionnaire validated to look at the health status of patients with a variety of forms of ILD. It consists of 15 items, and can be self-administered.

SECONDARY OUTCOMES:
MRC dyspnoea scale | 12 months
  A simple questionnaire quantifying the degree of dyspnoea suffered by patients, and shown to correlate well with direct measures of disability including walking distance, though is not quickly responsive to change

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Wilson, Principal Investigator — University of East Anglia
Locations (1):
- Norwich Medical School, Norwich, Norfolk, United Kingdom